# Resistance Testing Versus Adherence Support for Management of Virologic Failure on First-Line Antiretroviral Therapy in sub-Saharan Africa (REVAMP)

**Consent Forms** 

NCT 02787499

**Uganda and South Africa Versions** 

Version Date: 19th January 2018

# **Research Consent Form**

Protocol: Resistance Testing Versus Adherence Support for Management of Virologic Failure on First-Line Antiretroviral Therapy in sub-Saharan Africa

**Principal Investigator**: Dr. Yunus Moosa, University of KZN

**Co-Investigators:** Dr. Jaysingh Brijkumar; University of KZN

Dr. Pravi Moodley, University of UKZN

**Description of Subjects:** Patients with HIV currently on first-line ART with a detectable plasma viral load

>1,000copies/mL

Good day sir / madam

#### **Purpose**

We would like your permission to enroll you as a participant in a research study. Research is a process where investigators collect information on new ideas and study it to better understand what is going on. Your doctor has identified you as someone who is failing your first-line therapy for HIV. The research is aimed at understanding whether the current system of managing patients such as you who are failing treatment is preferred, or if additional blood tests will improve care.

#### **Procedures**

The study will include an initial visit and 2 or 3 additional visits (depending on the study group) spread out over the next 9 months. At each visit, we will collect information about you from your medical chart, such as test results and medications taken, and ask you some questions about your health. During each visit one or two tubes of blood will be collected (equivalent to 10 to 14 mL, or about 1 tablespoon). Also during certain study visits, a urine sample will be collected. We plan to enroll approximately 840 participants in the study. Half of them will be from South Africa and the other half from Uganda.

At today's visit, we randomly choose, like flipping a coin, which study group you will be in: half of participants will be randomly chosen for routine care with continued viral load monitoring and the other half will get an additional blood test immediately to see if they have resistance to their current treatments. Treatment and all medicines will continue to be provided to you by the clinic during the study, and will not be affected which group you are in. Those in the routine care group will return in 2-3 months for repeat viral load (or 1 month for pregnant women only), and again shortly thereafter to get their results and decide on the course of action, and then 6 months later for their final visit. Those in the resistance-testing arm will return when their resistance test results are back to decide on the course of action, and again about 9 months later to conclude the study. All participants will also be asked to keep their routine clinic appointments as recommended by their clinic providers. At the first visit, we will perform a pregnancy test for women of child bearing age (18 to 50 years old). Women who are pregnant and in the routine care group will be seen again at 1 month instead of at 2-3 months. We will also refer pregnant women to the antenatal care clinic, if they are not already enrolled. At each visit we will ask you some questions about your health, which will take no more than 30 minutes, and ask you to allow us to take your blood, which should take no more than 10 minutes. To draw your blood, the skin overlying a large vein of your forearm will be carefully cleaned with alcohol. A needle will then be inserted into the vein and, depending on the visit, 10 to 14 mL, or about 1 tablespoon of blood is withdrawn. During today's visit and the last visit, we will request that you to allow us to collect a urine sample for future tests. For those in the routine care group, we will also request that you allow us to collect a urine sample at the second visit, for future tests. Treatment will continue to be provided to you by the clinic during the study and will not be affected whether you do or do not take part in the study, or whether or not you withdraw during the study. Bloods and urine samples will be sent to Inkosi Albert Luthuli Central Hospital for testing. Urine samples will also be sent to UrSure, Inc in the United States for testing.

#### **Risks and Discomforts**

Blood drawing may cause a small amount of pain. In addition, a temporary bruise or "black and blue mark" may develop. Rarely, people faint after blood drawing. Very rarely, the vein in which the needle has been inserted may become inflamed or infected, which can be treated. There is the remote possibility that there could be a loss of confidentiality of your HIV status or other clinical information. At any time during the study, you will be provided the opportunity to discuss any concerns further with the study staff. Every effort will be made to minimize the risk for the above.

#### **Benefits**

You will be reimbursed for your time and effort at each visit, such that you will receive 50 Rand for every visit and 100 Rand for the final visit. You will receive viral load and resistance testing for free as part of the study. You may benefit from the additional viral load and resistance testing results, or the input from study clinicians trained in management of virologic failure. All ART regimens and other treatments will be provided by the HIV clinics. Finally, your involvement in this study may help study researchers and clinic partners understand how to best manage virologic failure in sub-Saharan Africa.

#### Alternatives/Voluntary Participation/Withdrawal

You will continue to receive treatment and medications from your care providers at the clinic whether or not you participate or withdraw from the study. Your participation in this study is voluntary. You are free to discontinue your participation in this study at any time without penalty or loss of benefits to which you are otherwise entitled. If you decide not to participate, your clinical care providers will continue to manage your disease based upon the highest of standards available. Should you wish to withdraw, notify your study staff or Dr. Yunus Moosa (see below) as early as possible in writing or verbally. Please allow a 7-day period to discuss your withdrawal to participation in the study with all the researchers. The study doctors have the right to discontinue your involvement in this study if it would be dangerous for you to continue, if you do not follow study procedures, if the investigator decides to end the study or for any other reason. You have the right to decline answering all or some of the questions in the questionnaire.

#### **Blood and Urine Storage**

For blood you donate now or if additional blood is donated in the future, some of that blood will be tested and some of that blood may be stored for future use. The urine collected at the study visits will also be stored for future use. These samples will be stored at Inkosi Albert Luthuli Central Hospital, and may be shipped to the United States for additional tests of medication levels or specialized HIV tests that are not available in South Africa. By signing this consent, you give permission to the investigators for this purpose. However, at any time you have the right to request that this blood and urine be destroyed and no further testing will be performed on it by contacting the researchers (see details below). Should you wish to withdraw all participation from this study (blood testing, urine collection, and questionnaire interviews) from the study, and the information already gathered will remain as part of the study and no further tests will be done on your stored blood and urine.

#### Confidentiality

Your information will be labeled with a code number that is unrelated to your medical record number. The link of your code to your name and medical record number will be kept in a locked filing cabinet in research offices at the University of KwaZulu-Natal. This information will be stored for 10 years. We will keep all information about you confidential. Only those people who are working on this research study or the Biomedical Research Ethics Committee will have access to this information. The doctors and counselors who normally treat you and are not part of the study will not have access to your questionnaire unless you request them to have access. You will not be personally identified by name in any presentation or publication resulting from this study. The data collected in this study and the stored samples of blood and urine may be used for other HIV-related studies as decided by the investigators. The BIOMEDICAL RESEARCH ETHICS COMMITTEE (BREC) will ensure that your samples are used for the correct tests. BREC will review all

protocols that will involve stored samples and approval will be obtained from BREC and consent from you before starting any new study.

### **Compensation / Costs**

You will be reimbursed 50 Rand at each study visit for your time and effort, until the final visit, for which you will receive 100 Rand for completion of the study. There will be no additional costs to you to participate in this study.

### **Study Contacts**

You can reach **Dr. Yunus Moosa** at **031 2604368** if you have questions, concerns or complaints about this study.

You can also reach the Biomedical Research Ethics Committee at **031 260 2486 or send fax to 031 260 4609 or send Email:** BREC@ukzn.ac.za if you have any questions about your participation.

#### **Entitlement**

You will receive a copy of this signed consent form for your records.

THIS RESEARCH HAS BEEN APPROVED BY THE BIOMEDICAL RESEARCH ETHICS COMMITTEE (BREC)

| SIGNATURES | |
|---|---|
| Subject | Date/Time |
| Subject's preferred contact information during course of st | udy: |
| I have explained the purpose of the research, the study prothe possible risks and discomforts and potential benefits. I research study to the best of my ability. | |
| Investigator/Individual Obtaining Consent | Date/Time |
| Witness | <br>Date/Time |

# Ifomu lokuvuma ukungena ocwaningweni

Protocol: Resistance Testing Versus Adherence Support for Management of Virologic Failure on First-

Line Antiretroviral Therapy in sub-Saharan Africa

Umcwaningi omkhulu: Dr. Yunus Moosa, University of KZN

**Ubalekeli babacwaningi:** Dr. Jaysingh Brijkumar; University of KZN

Dr. Pravi Moodley, University of UKZN

**Ukuchazwa kocwaningo**: Iziguli ezinakekelwa eMitholampilo yomphakathi yesandulela

ngculazi okuyiziguli ezingasetshenzelwa imishanguzo ngendlela

ukwehlisa inani lesandulela ngculazi egazini labo.

Sawubona

#### Inhloso

Sicela imvume kuwe yokuthi ubambe iqhaza ocwaningweni lwethu. Ucwaningo yinqubo lapho abacwaningi beqoqa khona ulwazi emiqondweni emisha bayicwaninge ukuze baqonde kangcono okwenzekayo. Uqokwe udokotela wakho njengomunye walabo abangasetshenzelwa imishanguzo esigabeni sokuqala yesandulela ngculazi. Ucwaningo kuhloswe ngalo ukuqonda ukuthi ngabe indlela esetshenziswa manje yokunakekela iziguli ezifana nawe ezingaphumeleli ohlelweni lokuqala lokwelashwa ingabe iyonayona na?

### Inqubo

Ulindeleke ukuba uvakashe izigaba ezintathu noma ngaphezulu (lokhu koya ngeqembu locwaningo ongene ngaphansi kwalo) Okuyokwenziwa ezinyangeni eziyisishaga lolunye. Ekuvakasheni ngakunye, siyothatha ulwazi lwakho kwi fayela lakho lezempilo, ulwazi olufana nemiphumela yokuhlolwa okwenzile kanye nemithi obuyithatha, bese sikubuza eminye imibuzo ngempilo yakho. Siyophinde ekuvakasheni ngakunye sithathe ishubhu noma amashubhu amabili egazi (alingana no 10 kuya ku 14 mL, noma elilingana nesipuni sokudla esisodwa) nesampula lomchamo ekuvakasheni kokuqala nokokugcina. Kulolucwaningo sihlela ukufaka abantu abalinganiselwa ku 840. Uhafu wabo baqhamuka e South Africa nomunye uhafu uqhamuka e Uganda.

Ekuvakasheni kwanamuhla sikhethe ngendlela yokuthi siphose imali phezulu okuyiyona ndlela esikhombisa ukuthi uzongena kuliphi iqembu: uhhafu wabazoba kulolucwaningo uyokhethelwa ukuqhubeka nokwelashwa nokuqhubeka nokubhekwa ubungako begciwane emzimbeni, omunye uhhafu kuyothathwa kuwo igazi ngalesosikhathi lihlolelwe ukubona ukuthi ngabe imithi abayisebenzisayo njengamanje ayiphikisani negazi lakho. Labo abaseqenjini lokwelashwa okujwayekile bayobuya ezinyangeni ezimbili kuya kwezintathu bazophinde bazohlolwa kubhekwa izinga legciwane egazini (noma inyanga eyodwa kulabo besifazane abakhulelwe kuphela), bese kuphinda ngemuva kwalokho babheke imiphumela okuyiyo eyolawula uhlelo okuyofanele balulandele emuva kwalokho, bese kuthi emuva kwezinyanga eziyisithupha beze ekuvakasheni kokugcina. Labo abaseqenjini elihlolelwa ukungasebenzi kwemishanguzo bayobuya uma imiphumela yabo seyibuyile nabo bathathe isinqumo sohlelo abazolulandela bese kuba sezinyangeni eziyisishagalolunye ukuzoqedela ucwaningo. Bonke abakulolucwaningo bayocelwa ukuthi bagcine ukuvakasha kwabo kwaseMtholampilo okulindelekile njengokuhlela kwabaseMtholampilo. Ekuvakasheni kokuqala, siyohlolela ukukhulelwa kubantu besifazane abaseminyakeni yokuthi bangakhulelwa (18 kuya ku eminyakeni ewu 50 ubudala). Abantu besifazane abakhulelwe futhi abaseqenjini elijwayelekile lokwelashwa bayobonwa futhi enyangeni yokuqala esikhundleni sasezinyangeni ezimbili kuya kwezintathu. Siyobuye sithumele abesifazane abakhulelwe eMtholampilo wabantu abakhulelwe uma bengakaze bawuqale uMtholampilo wabakhulelwe. Ekuvakasheni ngakunye siyokubuza imibuzo yezempilo okungeke kuthathe ngaphezu kwemizuzu engamashumi amathathu, siphinde sikucele ukuba usivumele sikhiphe kuwe igazi, nalokhu okungeke kuthathe ngaphezu kwemizuzu eyishumi. Ukuze sikhiphe kuwe igazi isikhumba esemboze umthambo omkhulu engalweni yakho siyohlanzwa ngokucophelela ngoketshezi lokuhlanza isikhumba. Inalithi iyofakwa emthanjeni kuyoya ngokuthi yikuphi lokhu kuvakasha kuyothathwa igazi elingeshubhu elilodwa noma amabili (elilingana no 10 kuya ku 14 mL, noma elingangesipuni sokudla). Kulokhu kuvakasha kwanamuhlanje nangokuvakasha kokugcina siyophinde sicele ukuba usivumele sithathe umchamo esiyowusebenzisa esikhathini esizayo. Uyoqhubeka nokuhlengwa kulomtholampilo ngesikhathi usekulolucwaningo futhi lokhu ngeke kuphazanyiswe wukuthi uyavuma yini noma awuvumi ukungena kulolucwaningo. Amasampula egazi nawomchamo ayothunyelwa esibhedlela e Inkosi Albert Luthuli Central Hospital ukuze ahlolwe. Amasampula omchamo ayophinde athunyelwe kwa UrSure, Inc eMelika ukuze ahlolwe.

#### Ubungozi kanye nokungaphatheki kahle

Ukukhishwa kwegazi kungabangela ubuhlungu obuncane. Ngaphezu kwalokhu, kungenzeka kuvele noma kube nomhuzukwana okwesikhashana noma umaka omnyama kanye nobuhlazana. Kuyenzeka nje ukuthi umuntu aquleke ngemuva kokukhipha igazi kepha akujwayelekile. Kuyenzeka futhi ukuthi umthambo lapho bekungene khona inalithi uvuvukale noma kubhibhe kepha lokhu kungelashwa. Kunethuba elincane kakhulu lokuthi ulwazi lokuthi uphila neSandulela Ngculazi kanye nemininingwane yakho yezempilo ingabi yimfihlo. Noma nini ngesikhathi kuqhubeka lolucwaningo uyoba nethuba lokukhuluma nabasebenza kulolucwaningo ngalokho okungakuphethe kahle kulolucwaningo. Kuyokwenziwa yonke imizamo ukunciphisa mathuba okuba kwenzeke noma yikuphi kulokhu okubalulwe ngenhla.

#### Inzuzo

Uyonxephezelwa ngesikhathi sakho nokuza eMtholampilo ngenxa yalolucwaningo. Uyonikwa U R50 ngokuvakasha ngakunye kuze kube ukuvakasha kokugcina, lapho uyonikwa khona u R100 uma uyofikela ukuzophetha ucwaningo. Uyonikwa imiphumela yokuhlolelwa ubungako begciwane emzimbeni wakho kanye nemiphumela yokuthi imithi ngabe iyakwazi yini ukulwisana negciwane emzimbeni wakho. Kungenzeka uhlomule ngokuba wenze okunye ukuhlolwa maqondana nobungako begciwane emzimbeni wakho kanye nokubheka ukuthi ngabe imithi ngabe iyakwazi yini ukulwisana negciwane emzimbeni wakho, noma ukwelulekwa ngabaqeqeshiwe kulolucwaningo abasebenza ukubheka ukungasebenzi kwemishanguzo ukwehlisa inani leSandulela Ngculazi egazini. Yonke ingxube yemishanguzo iyokhishwa uMtholampilo weSandulela Ngculazi. Ekugcineni, ukuba ungenele lolucwaningo kungasiza abacwaningi nabasebenzisana nabo eMtholampilo baqonde ukuthi bangasebenzisa ziphi izindlela ukubhekana nokuhluleka ukwehlisa inani lamagciwane eSandulela Ngculazi egazini e mazweni ase Africa.

# Ezinye izindlela/Ukungena ocwaningweni ngokuzithandela/Ukuphuma ocwaningweni

Uyoqhubeka welashwe futhi uthole imishanguzo eMtholampilo noma ngabe uyalungenela noma awulungeneli lolucwaningo. Ukungenela lolucwaningo kuwukuthanda kwakho awuphoqiwe. Wemukelekile ukuba uphume kulolucwaningo noma ingasiphi isikhathi ngaphandle kokujeziswa noma kokulahlekelwa amalungelo akho emtholampilo. Uma ukhetha ukungalungeneli lolucwaningo, udokotela okunakekelayo emtholampilo uyoqhubeka nokukunakekela ngayona yonke indlela ekhona. Uma usufisa ukuphuma kulolucwaningo, uyacelwa ukuba wazise osebenzisana nabo eMtholampilo noma wazise u Dr. Yunus Moosa ngokushesha ngokumbhalela noma ngomlomo (bheka ngezansi imininingwane). Sicela unike abacwaningi isikhathi esingangezinsuku eziyisikhombisa ukuthi sixoxisane ngokuphuma kwakho ocwaningweni. Udokotela wakulolucwaningo unelungelo lokukumisa ukuthi uqhubeke kulolucwaningo uma lokho kungabeka impilo yakho engozini, uma ungalandeli imigomo yalolucwaningo uma futhi umcwaningi ethatha isinqumo sokulumisa lolucwaningo nganoma ingasiphi isizathu. Unelungelo lokunqaba ukuphendula yonke imibuzo noma eminye imibuzo obuzwayona kulena ebhalwe phansi.

#### Ukugcinwa kwegazi nomchamo

Igazi onikela ngalo manje noma esikhathini esizayo elinye lalelogazi liyohlolwa elinye ligcinelwe ukusetshenziswa esikhathini esizayo. Umchamo oyothathwa ekuvakasheni kokuqala nokokugcina nawo uyogcinelwa ukusetshenziswa esikhathini esizayo. Lamasampula ayogcinwa e Inkosi Albert Luthuli Central Hospital, kungenzeka aphinde athunyelwe phesheya kwezilwandle e United States ukuze aphinde ahlolwe ngezindlela ezingekho lapha eNingizimu Africa. Ngokusayina lelifomu, unikeza abacwaningi lelogunya. Kepha, unelungelo lokuthi noma ingasiphi isikhathi ufune amasampula akho egazi nawomchamo achithwe

ngeke esasetshenziswa emuva kwalokhu uma ufuna ukuxhumana nabacwaningi (bheka imininingwane ngezansi). Uma ufuna ukuphuma kulolucwaningo ngokuphelele (ekuhlolweni kwegazi, ekuthathweni komchamo nokubuzwa kwemibuzo ebhalwe phansi), ulwazi oluvele seluqoqiwe luyogcinwa kulolucwaningo kepha ngeke kusaqhutshekwa nokusebenzisa amagazi nomchamo wakho ogciniwe.

#### **Imfihlo**

Ulwazi neminingwane yakho kuyofakwa inombolo ethile yakulolucwaningo engahambisani nemininingwane yakho yezempilo. Ukuxhumana okukhona phakathi kwe khodi negama lakho kanye nenombolo yakho yemininingwane yakho yezempilo kuyovalelwa emahovisi ocwaningo eNyuvesi yaKwaZulu-Natal. Lokhu kuyogcinwa iminyaka eyishumi. Siyogcina lonke ulwazi lwakho oluyimfihlo. Yilabo bantu abasebenza kulolucwaningo kuphela noma abekomidi locwaningo lase University (Biomedical Research Ethics Committee) abayokwazi ukufinyelela kulolulwazi. Odokotela abajwayele ukukwelapha kanye namakhansela abangeyona ingxenye yalolucwaningo angeke bakwazi ukufinyelela emininingwaneni yakho kanye nemibuzo yalolucwaningo, kuphela kungenzeka lokhu uma kusho wena. Angeke kubhalwe igama lakho kunoma yimiphi imibhalo eyimiphumela yalolucwaningo. Imininingwane eqoqwe kulolucwaningo namasampula egazi nawomchamo agciniwe angasetshenziswa abacwaningi kolunye ucwaningo lweSandulela Ngculazi ngendlela ababona ngayo. I BIOMEDICAL RESEARCH ETHICS COMMITTEE (BREC) iyoqinisekisa ukuthi amasampula akho asetshenziselwa ukuhlolwa okuyikhona. I BREC iyocubungula yonke imiqulu yocwaningo eyofaka ukugcinwa kwamasampula iphinde iphasise lemiqulu kutholakale nemvume kozoba kulolucwaningo ngaphambi kokuba kuqale noma yiluphi ucwaningo olusha.

#### Isinxephezelo / Izindleko

Uyobuyiselwa imali engu R50 ekuvakasheni ngakunye ngesikhathi sakho nokuzama ukuza ocwaningweni kuze kube ukuvakasha kokugcina lapho uyothola khona u R100. Azikho ezinye izindleko oyobhekana nazo.

#### Imininingwane vokuxhumana noMcwaningi okhulu

Ungaxhumana no **Dr. Yunus Moosa ku 031 2604368 uma unemibuzo noma kukhona ongenamile ngakho ngalolucwaningo**.

Ungaxhumana futhi ne Biomedical Research Ethics Committee ku **031 260 2486 noma uthumele** isikhahlamezi ku **031 260 4609 noma uthumele umyalezo ngekhompyutha / Email: BREC@ukzn.ac.za** uma uba nemibuzo ngokuba kulolucwaningo.

#### Okuyilungelo lakho

Uyothola ikhophi yalelifomu olisayinile kulolucwaningo ukuze uzigcinele lona.

LOLUCWANINGO LUPHASISIWE YI KOMIDI LOCWANINGO I BIOMEDICAL RESEARCH ETHICS COMMITTEE (BREC)

| AMASIGINESHA | | |
|---|---|---|
| Okwenziwa ngaye ucwaningo | Usuku/isikhathi | |
| Imininingwane yokuxhumana emini nokwenziwa ngaye ucwaningo: | | |
| | | - |

Ngiyichazile inhloso yalolucwaningo, nezinqubo zakhona, ngachaza lezo eziwucwaningo, nobungozi balolucwaningo nokungenzeka kungmphathi kahle okwenziwa ngaye ucwaningo kanye nalokho okungaba yinzuzo kuye. Ngiphendulo yonke imibuzo ngalolucwaningo ngokusemandleni ami onke.

| Umcwaningi/Othole imvume kokwenziwa ngaye ucwaningo | Usuku/isikhathi |
|-----------------------------------------------------|---------------------|
| Ufakazi | <br>Usuku/isikhathi |

# MBARARA UNIVERSITY OF SCIENCE AND TECHNOLOGY RESEARCH ETHICS COMMITTEE

P.O. Box 1410, Mbarara, Uganda

Tel: 256-4854-33795 Fax: 256 4854 20782

Email: <u>irc@must.ac.ug</u> <u>mustirb@gmail.com</u>

Web site: www.must.ac.ug



#### INFORMED CONSENT DOCUMENT

**Study Title:** 

REVAMP Study [Resistance Testing Versus Adherence Support for Management of Patients with Virologic Failure on First-Line Antiretroviral Therapy in sub-Saharan Africa]

Principal Investigator(s): Dr. Bosco Mwebesa Bwana, Dr. Mark Siedner

#### INTRODUCTION

The main goal of treating HIV with antiretroviral drugs is to control the HIV virus, improve health of those who are infected and prevent transmission. However, rates of treatment failure for people with HIV taking antiretroviral therapy are high. The overall goal of this study is to see if it is possible to improve care of patients with HIV and treatment failure in sub-Saharan Africa, and if so, if it can be done in a way that is affordable to patients and the healthcare system. The research is being lead by in Uganda by Dr. Bosco Bwana of Mbarara University of Science and Technology, and Dr. Mark Siedner of the Massachusetts General Hospital.

### What you should know about this study:

- You are being asked to join a research study.
- This consent form explains the research study and your part in the study
- Please read it carefully and take as much time as you need
- You are a volunteer. You can choose not to take part, and if you join, you may quit at any time. There will be no penalty if you decide to quit the study

#### **Background**

Approximately 1 in 3 patients with HIV infection in sub-Saharan Africa taking antiretroviral therapy will fail therapy and have the virus return in their blood within two years of starting treatment. The current recommendations for monitoring of patients who have failed therapy is to offer adherence counseling, repeat testing for virus in the blood in 3-6 months, and then decide if drugs should be changed. However, it is not known if adding a second test, called a resistance test, to see if the virus has changed in ways to make drugs less effective, will improve care of patients and avoid unnecessary switching of drugs to more expensive second line regimens. This study aims to see if additional tests will have a beneficial impact on treatment of patients with HIV who have failed therapy.

### Purpose of the research project:

The purpose of this study is to see whether the current system of managing HIV patients with treatment failure is optimal, or if a second test can help improve care. We are expecting to study approximately 420 patients in Uganda and 420 patients in South Africa in this project. Half of the patients enrolled will be randomly selected to get the current standard of care, and the other half will get a second test to see if it improves patient health. Study participants will remain in the study for approximately 9 months.

# Why you are being asked to participate:

You are being asked to participate in this study because you are an adult with HIV infection, taking antiretroviral therapy and actively in care at the clinic, but have detectable virus in your blood suggesting treatment failure.

#### **Procedures:**

For those who agree to be part of the study, they will be divided into one of two groups after completing the informed consent process. You will be assigned by chance, like the flip of a coin, into one of two groups:

- 1) Group One (standard care): Study participants in the first group will continue with the standard of HIV care. They will receive adherence counseling today, a repeat blood test to check for the HIV virus again in 2-3 months (or 1 month for pregnant women only), and then meet with study and clinic staff when the result is ready to decide if their HIV drugs should be changed or remain the same. They will be seen by study staff for one final visit approximately nine months from now to check their blood one last time to see if the virus is still present or under control. They will continue with their normal clinic schedule and procedures in the meantime and after the study ends.
- 2) Group Two (resistance testing): Study participants in the second group will get another blood test today to see if the virus in their blood has resistance to drugs. They will return as soon as the result is ready and meet with study and clinic staff to decide if their HIV drugs should change or remain the same. They will be seen again by study staff in approximately nine months to check their blood one last time to see if the virus is still present or under control. They will continue with their normal clinic schedule and procedures in the meantime and after the study ends.

This study will last approximately 9 months and include three (Group One) or two (Group Two) additional study visits after today. If you agree to participate in the study you will be asked to complete the following procedures:

- 1. **Interviews**: We will ask you about your health, what medical care you have received recently, and your history of treatment with HIV infection. We will also ask you about your quality of life and whether you feel content and healthy. We will ask you these questions to see if the procedures in the study have a beneficial impact on the quality of life for people with HIV infection. The interview will take approximately 30 minutes to complete.
- 2. **Record Review**: Study staff will ask the clinic staff for access to review your medical records. This review will include your dates of diagnosis of HIV, when you began to receive care at the clinic, the medicines you have received, and the medical problems or drug side effects you have had. This information will help us understand how the interventions received in the study affect your health, your treatment, and the costs of healthcare.
- 3. **Blood tests**: We will draw your blood at each study visit. The total amount of blood to be drawn will be no more than three tubes (15cc, or 3 teaspoons) on any given day, and no more than five tubes (40cc, or 8 teaspoons) over the total study duration. The blood tests will be used to test the levels of HIV virus in your blood and whether the antiretroviral therapy drugs you take are effective at killing the virus. We will also be storing your blood to do tests of your blood later for levels of the virus, drug resistance, and to check the level of antiretroviral drugs in your blood at a later date.

- 4. Phone and Home Tracking: If you miss your study visit or do not show up, we will try and contact you to remind of your visit and encourage you to return to complete the study. If we cannot get a hold of you by phone, we may try and find you at your home to prompt to you to return to care and complete the study. The study staff will call to attempt to notify you before conducting home visits.
- 5. **Pregnancy test.** If you are a woman under the age of 50, you will take a urine pregnancy test when you are enrolled in the study. If you are found to be pregnant, and in the standard care group (group 1), you will be seen again at 1 month instead of at 3 months. We will also be sure you are referred to the antenatal care clinic, if you are not already enrolled.
- 6. **Urine tests.** Each time we collect blood for study purposes, we will also request a urine sample for collection. We will store your urine to do tests to check the level of antiretroviral drugs in your urine at a later date. Because these tests will be done later, results will not be available to share with you.

#### Risks / discomforts:

- 1. You may feel uncomfortable that data about your health is being shared with researchers. We will make every effort to protect your privacy. Any paper forms used as part of this study will be stored in a locked file cabinet that remains in a locked study office. All other records will be stored in a password-protected database in the United States. Aside from this consent form and a single address form, all other study documents will only identify you with a coded identification number and only trained research staff and study team members will have access to the data.
- 2. Allowing research assistants or other study staff to come to your home to find you for study visits or collect samples may result in members of your family or community knowing that you are participating in the study. No study team members will visit you unless you are missing from your appointments. In the event a study team member does visit, they will only do so after trying to arrange a convenient time for you and will do so in unmarked vehicles.
- **3.** There is the risk of discomfort when your blood is drawn. There is also a small risk of bruising or infection. We will minimize this risk with the use of experienced and trained phlebotomists. No more than 3 teaspoons of blood will be drawn on any day.

# **Sharing of research records**

Your research records may be shared confidentially among investigators who are working with Drs. Siedner and Bwana on this study. They are located at Mbarara University, Uganda and the Massachusetts General Hospital/Harvard University, USA. Your research results may also be shared, without any information about your personal identity, with governmental health research databases of genetic information. These data include data from the clinic database. You may decline permission to share your records at any time. Any request that your records not be shared should be made either in writing or verbally to the study staff. Such requests will be honored for future research, but data that have already been distributed to researchers cannot be retracted. Your research records will not be sold, but may be used to develop useful drugs or medical tests.

#### **Benefits:**

You will receive results of the pregnancy test (if eligible) and blood tests, including results of HIV viral load tests and HIV antiretroviral therapy resistance tests. All study participants will also receive results of their tests (viral load and resistance tests) after the final study visit in about 9 months. A member of the study staff will contact you when the blood test results are done and to arrange a time that you can return for your next visit and/or collect the results. These tests might help identify changes in your HIV treatment that are recommended by clinic staff. While there may be no direct benefit to you by participating in the study, there may be benefits to the public through the understanding of how to best manage patients with HIV.

# Incentives / rewards for participating:

You will be reimbursed for your transportation costs home from the study site on the day of enrollment and future study visits. The amount of the reimbursement will be determined based on your distance from clinic (range 10,000 – 30,000 Ugandan Shillings). You will also be given a bar of soap or a kilogram of sugar to compensate you for your time. The costs of viral load and resistance testing performed as part of this study will be covered by the study, and we will provide results of these tests to you and your clinicians to help ensure you receive appropriate care, including any changes to your HIV medicines, in response to these results. The study itself will not provide medications or compensation for medicines, but we will refer you to the clinic to receive them.

#### **Protecting data confidentiality:**

Participation in research can involve a loss of privacy. Your research records will be handled as confidentially as possible. All research records will be coded so that no person outside the study group can identify you. No individual identities will be used in any reports or publications that result from this study. No individual identities will be included in genetic data shared with other researchers. Your doctor will not have access to any of the information you give the researchers, unless you give the study your consent to share your laboratory results.

# Protecting subject privacy during data collection:

All interviews will be conducted in a private place, the research assistant will help protect your privacy by not discussing your responses with anyone else.

#### Right to refuse / withdraw:

You may choose to not participate without the risk of losing your current healthcare or medicines. To do so you only need to inform the study staff of your intention to withdraw either verbally or in writing.

# What happens if you leave the study?

You can choose at any time not to take part in the study. There will be no penalty to you for doing so and you will resume standard care at your treatment clinic.

# Who do I ask/call if I have questions or a problem?

If you have any additional questions, you can call the Principal Investigator, Dr. Bosco Bwana at 0772308895. If you have questions for the Institutional Ethical Review Committee at Mbarara University, you can call Dr. Francis Bajunirwe at 0485433795 or write to MUST- IRC P.O BOX 1410 Mbarara, Uganda

#### Contact for IRC office

Dr. Francis Bajunirwe Chairman MUST-IRC P.O Box 1410 Mbarara Tel: 0485433795

#### Consent

You have been given a copy of this consent document.

PARTICIPATING IN THIS STUDY IS VOLUNTARY

You have the right to withdraw at any time without affecting your care.

# What does your signature (or thumbprint/mark) on this consent form mean?

Your signature on this form means

- You have been informed about this study's purpose, procedures, possible benefits and risks
- You have been given the chance to ask questions before you sign
- You have voluntarily agreed to be in this study

| Print name of adult participant | Signature of adult participant/legally Authorized representative | Date |
|---|---|---|
| Print name of person obtaining Consent | Signature | —<br>Date |
| Print name of witness | Signature of witness | <br>Date |

# MBARARA UNIVERSITY OF SCIENCE AND TECHNOLOGY RESEARCH ETHICS COMMITTEE

P.O. Box 1410, Mbarara, Uganda

Tel: 256-4854-33795 Fax: 256 4854 20782

Email: <u>irc@must.ac.ug</u> <u>mustirb@gmail.com</u>
Web site : <u>www.must.ac.ug</u>



#### EKIHANDIIKO KY'OKUSHABA KWEJUMBA OMUMUSHOMO

#### **OMUTWE GW'OMUSHOMO:**

ENKORA ENSTYA: Okugyeragyeranisa oku omubiri gurikwanga omubazi hamwe n'okubangirwa kuhamira ahamibazi eyokujanjaba abarweire ab'akakooko ka sirimu abu kagumire nikeyongyera omushagama obwe bari aha kika ky'okubanza ky'emibazi emihango omumashuuma ga Africa.

ABACONDOZA ABAKURU: Dr. Bosco Mwebesa Bwana, Dr. Mark Siedner

#### **OKWANJURA**

Ekigyendererwa ekikuru eky'okujanjaba akakooko ka sirimu n'emibazi emihango (ARVs) n'okutanga akakooko kasirimu, kwongyera kushemeza amagara gaabo abarweire kandi n'okuremesa okujanjaara. Kwonka, okuremwa omukujanjaba abarweire bakakooko ka sirimu abarikumira emibazi emihango kuri aheiguru. Ekigyendererwa ekikuru ekyomushomo ogu nokureeba kyaba nikibasika kutunguura obujanjabi bwabarweire bakakooko ka siriimu hamwe nabaremirwe obujanjabi omumashuma ga Africa, kandi kyaba kiri ekyo, kyaba nikibasiika kukorwa omungyeri ekubasiika omubya sente ah'abarweire hamwe n'enkora y'obujanjabi. Okucondoza nikwebemberwa omu Uganda Dr. Bosco Bwana owa Mbarara University of Science and Technology, hamwe na Dr. Mark Siedner owa Massachusetts General Hospital

### Ekyoshemereire kumanya ahamushomo ogu:

- Oriyo n'oshabwa kwejumba omumushomo gw'okucondoza.
- Ekihandiiko ky'okushaba okwejumba eki nikikushoborera omushomo hamwe n'omwoga gwawe omumushomo ogu.
- Nyabura shoma orikwetwara kandi otware obwire bw'okwetaga bwoona.
- Ori nyekundiire. Nobaasa kusharamu obutejumba, kandi k'orayejumbe, obaasa kuruga omumushomo eshaha yoona. Tiharabeho kibonerezo k'orasharemu kuruga omumushomo.

#### Oburugo bw'omushomo

Omurweire nka 1 ahari 3 abeine akakooko ka sirimu omumashuuma ga Africa abakumira ARVs nibaza kuremwa obujanjabi kandi kiretere akakooko kagaruka omushagama yaabo omumyaka 2 yokutandiika obujanjabi. Obuhabuzi oburikuhebwa obwahati bw'okurebuuza obarweire abaremirwe obujanjabi n'okuhereza okuhumurizibwa omu by'okugumizamu omubazi, kugarukamu okucebera obukooko omushagama omumyezi 3-6, kandi hakakorwa okusharamu yaaba emibazi eshemereire kuhindurwa. Kwonka, tikirikumanywa yaba okwongyeraho okucebera kwakabiri okurikureba yaba akakooko kahindwirwe omumitwarize kwangira okukora kw'omubazi (resistance test), kibaasa kutunguura obujanjabi bw'abarweire kandi tuketantara okuhindura emibazi yekika kya kabiri okuteine ekigyendererwa kandi ekirikusera omubyasente. Omushomo ogu gw'orekyereire kureeba yaba okucebera okurikwongyerwaho kubaasa kureta empinduka enungi aha kujanjaba abarweire bakakokok ka sirimu abaremirwe obujanjabi.

### Ekigyendererwa ky'omushomo:

Ekigyendererwa kyomushomo ogu n'okureba yaba enkora eriho obwahati eyo kujanjaba abarweire bakakooko ka sirimu abaremirwe emibazi n'emara, nari okucebera okwa kabiri kukwakubaasa kuyamba kutungura obujanjabi. Turiyo nitutebereza kushoma ahabarweire nka 420 omu Uganda hamwe na 420 omw'eihanga rya South Afrika omumushomo ogu. Ekicweka kyabarweire nikiza kutoranirwa eryo kutunga enkora ey'obujanjabi eriho obwahati, kandi ekicweka ekindi nikiza kutunga okuceberwa okwa kabiri kureba yaba nikuza kutunguura amagara g'omurweire. Abayejumba babaasa kumara omumushomo emyezi nka mwenda.

### Ahabwenki n'oshabwa kwejumba:

Oriyo n'oshabwa kwejumba omumushomo ogu ahakuba ori omuntu mukuru oyine akakooko ka sirimu, nomira emibazi emihango kandi notunga obujanjabi aheirwariro eri, kwonka obukooko bwasirimu nibukirebeka omushagama yawe ekirikworeka ngu oremirwe obujanjabi.

#### Entwaza:

Abarikirize kwejumba omumushomo ogu, nibaza kubaganisibwamu omu bibiina/guruupu ibiri bwanyima y'okuhendera ekikorwa ky'okushaba kwejumba omumushomo. Nituza kutoranira eryo omuntu kuza omu guruupu egi nari endijo:

- 3) <u>Guruupu 1 (obujanjabi obwaburijo</u>): Abejumbire omu guruupu 1 nibaza kugumizamu nobujanjabi bw'akakooko ka sirimu obwaburijo. Nibaza kuhumurizibwa omuby'okuguma ahamubazi erizooba, nibaza kugaruka baceberwe eshagama kureeba akakooko omu myezi 2-3 (nari omwezi 1 ahabw'abakazi b'enda bonka), kandi babugane abakozi b'omushomo hamwe n'eirwariro ebirugamu byaheza kumanywa kugira ngu okusharamu kukorwe yaba emibazi y'akakooko ehindurwe nari ogume n'egyo. Nibaza kureebwa abakozi bomushomo ahabw'orutayayo rw'ahamuheru (Emyezi mwenda kuruga hati) kucebera eshagama omurundi gumwe gwahamuheru kureeba akakooko kaba kakirimu nari katangirwe. Nibaza kugumizamu nenkora yeirwariro eyaburijo hamwe n'entwaza kandi bwanyima omushomo guhwe.
- 4) <u>Guruupu 2</u>: Abejumbire omumushomo omu guruupu ya kabiri nibaza kutunga okuceberwa eshagama okundi erizooba kureeba yaba akakooko omushagama yaabo nikangira emibazi. Nibaza kugaruka ebyaruga omukucebera byabo byaheza kumanywa kandi babugane abakozi b'omushomo hamwe n'eirwariro ebirugamu byaheza kumanywa kugira ngu okusharamu kukorwe yaba emibazi yakakooko ehindurwe nari ogume n'egyo. Nibaza kurebwa abakozi bomushomo ogundi nk'amezi mwenda kucebera eshagama ogundi murundi kureeba yaba akakooko kaba kakirimu nari katangirwe. Nibaza kugumizamu nenkora yeirwariro eyaburijo hamwe n'entwaza kandi bwanyima omushomo guhwe.

Omushomo ogu niguza kumara nk'emyezi 9 kandi habeho entayayo ezindi 3 (guruupu 1) nari 2 (guruupu 2) bwanyima y'erizooba. K'orabe noyikiriza kwejumba omumushomo ogu noza kushabwa kumarira entwaza ezi:

- 7. **Okubuuzibwa**: Nitwija kukubuuza aha magara gaawe, obujanjabi obwotungirenenyimaho, kandi n'ebyafaayo byawe ahakuraguza akakooko ka sirimu. Kandi nabwo nitwija kukubuuza amagara gorikutuura hamwe na waaba nohurira gye kandi omazirwe. Nitwija kukubuuza ebibuuzo ebi kureeba yaba entwaza z'omushomo zibiire ezomugasho ahamagara g'abantu abeine akakooko kasirimu. Okubuziibwa nikuza kutwara edakiika nka 30 kuhwa.
- 8. **Okureeba aha kipande**: Abakozi b'omushomo nibaza kukushaba abakozi beirwariro kureeba aha bipande byaawe. Eki kirimu okureeba ebiro by'okuceberwa akakooko ka sirimu, obw'obaanza kutunga obujanjabi aheirwariro, emibazi y'otungire, hamwe n'obuzibu

bw'omubazi obw'otungire. Amakuru aga nigaza kutuhwera kwetegyereza okw'enkora z'omushomo zihindwire amagara gaawe, obujanjabi hamwe n'enshohoza aha kuraguza.

- 9. Okucebera eshagama: Nituza kukwihaho eshagama buri rutayayo rw'omushomo. Eshagama erakwihweho yoona teraregye bucupa 3 (15cc, nari obugiko bwa sukari 3) omwizooba rimwe, kandi butakurenga obucupa 5 (40cc, nari obugiiko bwa shukari 8) omumushomo gwoona. Okucebera kweshagama nikuza kukozesibwa kupima obwingi bwakakooko omushagama yaawe hamwe nayaba emibazi emihaango eyokumira nebwita kurungi. Kandi nituza kuba nitubiika eshagama yaawe kucebera obwingi bwakakooko bwanyima, ahabw'obwingyi bwakakoko, okwanga kwomubazi, hamwe n'obwingi bw'omubazi omubiro ebyokwija.
- 10. Amasiimu hamwe n'okukuratiriza omuka: K'orayoshe orutayayo nari wabura kureebeka, nituza kugyezaho kukuhikirira kukwijutsya orutayayo rwawe kandi tukugaruzemu amaani gokweija okahendera omushomo. Twabura kukutunga ahasimu, nituza kugyezaho kandi tukushange omuka kukwijutsya kugaruka ahabujanjabi hamwe n'omushomo.
- 11. **Okucebera enda.** Waba ori omukazi ori ahansi y'emyaka 50, noza kuceberwa enkari kureeba yaba oyine enda waba otahibwe omumushomo. Washangwa oyine enda, kandi ori omu guruupu eyobujanjabi obwa burijo (guruupu 1), noza kureebwa ogundi murundi bwanyima y'omwezi 1 omumwanya gwa 3. Nituza kureebeka ngu wayehorezibwa omu karwariro akokureberera abakazi b'enda, beitu waba otakagireyo.
- 12. **Okucebera enkari.** Buri kukwihaho eshagama y'okucebera ahabw'omushomo, nikuza kukushaba ngu otuhe n'enkari y'okucebera. Nituza kubiika enkari yaawe kucebera kureeba orwingano rw'emibazi yakakooko ka sirimu omunkari yaawe omubiro eby'omumeisho. Ahakuba okucebera oku nikuza kukorwa nyetsya, ebyarugamu tibirabeho kubaganwa neiwe.

# Ebihikirizi/Ebyakukubuza obusingye:

- 4. Obaasa okugwibwa kubi kugira ngu ebirikukwata aha magara gaawe biriyo nibibaganwa n'abacondoza. Nituza kukora ekirikubasika kukuma ekihama kyawe. Empapura zirakozesibwe omumushomo ogu niziza kubikwa omu shandukye y'ekyoma erikuguma esibire omu ofisi y'omushomo. Ebihandiiko ebindi nibiza kubiikwa ahamikutu ya karimagyezi ekumirwe n'obunamba bw'ekihama omu Amerika. Oyihireho ekihandiko ky'okushaba kwejumba hamwe n'ekyendangiriro y'owawe, ebindi bihandiiko by'omushomo nibiza kutebwaho enamba z'ekihama kandi abakozi bomushomo abatendekirwe boonka nibo bararebe amakuru ago.
- 5. Okwikiriza abokuhwera omukucondoza nari abandi bakozi bomushomo kwija omuka yaawe ahabw'entayayo z'omushomo nari kwakiira eby'okucebera kubaasa kuretera abeka yaawe nari abekyanga kumanya ngu n'oyejumba omumushomo. Tihine muntu weena owomushomo arakutayayire kureka wabura ahantayayo. Omukozi w'omushomo yakutayayira, nibaza kukikora bwanyima y'okutebekanisa obwire burungi kandi nikiza kukorwa namotoka zitine bihandiiko.
- **6.** Hariho ekihikirizi ky'okuhurira kubi eshagama yaba n'ekwihwaho. Hariho akahiirizi kakye kokufuruta nari kushasha. Nituza kukyendeza ekihikirizi eki nabakoozi batendekirwe. Obujiiko bwa shukari butakurenga 3 bw'eshagaama nibuza kukwihwaho omwizooba.

# Okubagana ebihandiiko by'omushomo

Ebihandiiko byawe by'omushomo bibaasa kubaganwa omungyeri y'ekihama omubacondoza abakukora na abashaho Drs. Siedner and Bwana aha mushomo ogu. Nibashangwa ahari Mbarara University, Uganda hamwe n'ahairwariro erihango erya Massachusetts General Hospital/Harvard University, Amerika. Ebyaruga omu kucondoza bitariho ndanga muntu zaawe bibaasa kubaganwa namabikiro g'ebyokucondoza aga gavumenti. Amakuru aga garimu ebyihwa omumabikiro g'eirwariro. Obaasa kwanga obutabagana ebikukukwataho eshaha yoona. Okushaba kwoona kugira ngu amakuru gakukukwtaho gatabaganwa kushemereire kukorwa omu bigambo nari omubuhandikye aha bakozi b'omushomo. Okushaba nkokwo nkuza kutebwamu ekitinisa ahabw'okucondoza kwa nyetsya, kwonka amakuru agaheirwe abacondoza tigakeihwayo. Amakuru g'ebyokucondoza tigaraguzibwe, kwonka nigaza kukozesibwa kukora emibazi y'omugasho nari okucebera.

#### Amagoba:

Noza kutunga ebyaruga omu kucebera enda (waba otahire omumushomo hamwe nebyaruga omushagama, obariremu ebyaruga omukucebera obwingi bwakakooko hamwe n'oku akakooko karikwangira omibazi. Abejumbire omumushomo boona nibaza kutunga ebyaruga omukucebera (obwingyi bw'akakooko hamwe n'okwakakooko kakwangira emibazi) bwanyima y'orutayayo rw'ahamuheru omu myezi nka mwenda. Omwe ahabakozi b'omushomo nibija kukuhikirira eby'okucebera byaheza kurugamu kandi n'okukutebekanisiza obwire bworagarukye aharutayayo orundi kandi/ nari okakira obyarugamu. Okucebera oku kubaasa kuyamba kureeba empinduka omu bujanjabi bwawe bw'akakooko ka sirimu oburahebwe abakozi b'eirwariro. Nobuharabe habaasa kubura amagoba gahonaho ahabw'okwejumba omumushomo, habaasa kubaho okuganyirwamu omubantu ahabw'okwetegyereza okwabarweire b'akakooko ka sirimu babaasa kujanjabwa.

#### Okushumbusha/ ebirabo ahabw'okwejumba:

Noza kushashurwa enshohoza yawe ahabyentambura kuruga ahamwanya gw'omushomo kuza omuka ahizooba ry'okutaha omumushomo hamwe n'entayayo z'omushomo eza nyetsya. Omuhendo gw'okushumbusha niguza kurugirira rugyendo rwawe okurukwingana kuruga ah'eirwariro (kwiha ahari Shs 10,000 – 30,000 eza Uganda). Noza kuhebwa n'omuti gwa sabuuni nari kilo ya sukari kushumbusha obwire bwaawe. Esente z'okushashura okucebera obwingyi bw'akakooko hamwe n'okakwangira emibazi kwak'akakooko okurakorwe omumushomo neza kushashurwa omushomo. Torashashurwe ahaw'okuraguza okurakugambirwe kutunga ahabwebyarugamu obwo oyejumbire omumushomo ogu, nituza kukuha ebyaruga omukucebera kandi abashaho baawe nibeija kukuhwera kutunga obujanjabi obuhikire, obariremu n'okuhindura ahamibazi y'akakooko, kurugirira okwebirugamu biri. Omushomo tigwegurakuhereze emibazi nari enshohoza aha'mibazi, kwonka nituza kukwehoreza ah'eirwariro kubitunga.

# Okukuma ebihama by'amakuru:

Okwejumba omumushomo kibaasa kubamu ebihama byawe kushohora. Ebihandiiko by'okucondoza byawe nibiza kubiikwa nk'ekihama nk'okukikubasika. Ebihandiiko byawe by'okucondoza nibiza kuhebwa enamba kugira ngu tihine muntu aheru y'omushomo abaasa kukumanya. Tihine ndanga muntu eziratebwe ahamakuru gaawe agarashohozebwe ahamikutu yamakuru. Tihine ndanga muntu eziratekwe ahamakuru agarabaganwe n'abandi bacondoza. Omushaho waawe taratungye amakuru goona ag'orahe abacondoza, kwihaho wahereza omushomo orusa ngu babagane ebyaruga omukucebera.

# Okukuuma ekihama ky'owayejumba omukurundana amakuru:

Okubuzibwa kwoona nikuza kukorerwa omumwanya gwehereire, omuhwezi wokucondoza naza kukuma ekihama kyawe obwe atakuganira ebigarukwamu n'ondijo muntu.

# Obugabe bw'okwanga / kurugamu:

Obaasa kusharamu obutejumba kandi hatabireho ekihikirizi ky'okuferwa obujanjabi nari omubazi. Kukora ekyo noyetaga kumanyisa omukozi w'omushomo kwogyendereire kuruga omumushomo omubigambo nari omubuhandikye.

# Nihabahoki naruga omumushomo?

Obaasa kusharamu eshaha yoona obutejumba omumushomo ogu. Tiharabeho kibonererezo ahabwokukora ekyo kandi noza kugaruka ahabujanjabi obwa burijo ah'eirwariro.

#### Nimbuuza oha naba nyine ebibuuzo nari obuzibu?

K'orabe oyine ebibuuzo bikweyongyeraho, nobaasa kuterera omucondoza omukuru, Dr. Bosco Bwana ahari 0772308895. K'orabe oyine ebibuuzo byakakiiko k'entwaza n'emicwe y'ebyokucondoza ahari Mbarara University, nobaasa kuterera Dr. Francis Bajunirwe ahari 0485433795 nari ohandikire MUST- IRC P.O BOX 1410 Mbarara, Uganda

# Endagiriro ya ofisi IRC

Dr. Francis Bajunirwe Chairman MUST-IRC P.O Box 1410 Mbarara

Tel: 0485433795

#### Okushaba

Wahebwa kopi y'ekihandiiko ky'okushaba eki.

#### OKWEJUMBA OMUMUSHOMO OGU NINYEKUNDIRE

Oyine obugabe kurugamu eshaha yoona hatine kihindukire ahabujanjabi bwawe.

#### Omukono gwaawe (nari ekinkumu) ahakihandiiko ky'okushaba eki nikimanyisa ki?

Omukono gwawe ahakihandiiko nikimanyisa

- Wamanyisibwa ahabigyendererwa, entwaza, amagooba n'ebihikirizi by'omushomo.
- Wahebwa omugisha kubuuza ebibuuzo otakatireho omukono
- Wayekundira kwejumba omumushomo ogu

| Eiziina ry'owayejumba omukuru | Omukono gw'owayejumba omukuru/<br>Omuntu okwikirizibwa kujwekyera | Ebiro |
|---|---|---|
| Eiziina ry'ookushaba okwejumba | Omukono gw'owashaba kwejumba | _<br>Ebiro |
| Eiziina rya kareebi | Omukono gwa kareebi | Ebiro |